CLINICAL TRIAL: NCT03060421
Title: Evaluation of the Safety of Intraarticular Aquamid Reconstruction Injection for Knee Osteoarthritis in Humans
Status: Completed | Type: Observational
Sponsor: Henning Bliddal (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: P142.0
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Aquamid Reconstruction: Patients that have been treated with at least one intra-articular injection of aquamid as a treatment of osteoarthritis of the knee
  Interventions: Device: Aquamid reconstruction

INTERVENTIONS:
Device: Aquamid reconstruction — Aquamid Reconstruction is a Polyacrylamide hydrogel that contains 2.5% polyacrylamide and 97.5% non-pyrogenic water, with a unique molecular structure that allows the normal water exchange with the surrounding tissue without losing shape. Aquamid Reconstruction is biocompatible, non-absorbable non-biodegradable, stable, and sterile. T Aquamid Reconstruction is injected into the knee joint cavity.

SUMMARY:
As the use of Aquamid Reconstruction as an intraarticular device on humans is a relatively novel treatment, it is relevant to assess the safety profile of the device in a safety study to evaluate the safety of the device.

This is a retrospective single center cohort study of patients with osteoarthritis of the knee(s) that have been treated for knee OA referred to a clinical evaluation at our department.

The study consists of one clinical visit, at which the patients medical history will be taken and upon informed consent adverse events data is collected from medical records.

The study is retrospective.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated with intra-articular Aquamid Reconstruction in the knee for knee osteoarthritis and referred to our clinic for evaluatino of possible adverse device events.

Exclusion Criteria:

- There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 161 participants the total number of patients treated for Knee OA with Aquamid Reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Adverse Device Events | Day 1 (at the clinical examination)
  The investigator will examine each participant for evidence of adverse device events (ADEs) retrospectively by review of medical records and participant interview, and currently by a clinical examination

OTHER OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Day 1 (at the clinical examination)
  The WOMAC is a patient reported questionnaire that is easy to use and evaluates three domains; pain (five questions), stiffness (two questions) and physical function (17 questions), each weighted on a similar computation. The WOMAC Index is sensitive to change and is valid for elderly subjects with knee OA.
  To obtain the WOMAC scores, we apply the Knee Injury and Osteoarthritis Outcome Score (KOOS). The KOOS includes WOMAC Osteoarthritis Index LK 3.0 in its complete and original format (with permission), and WOMAC scores can be calculated (how to calculate WOMAC scores is presented in the document "KOOS scoring", available from www.koos.nu).
Knee joint range of motion | Day 1 (at the clinical examination)
  A clinical evaulation of knee joint range of motion. Will scored as 'normal' or 'reduced'
Global perceived effect of treatment | Day 1 (at the clinical examination)
  The participants will also answer a transition questionnaire on which the participants initially answers if their current state is "unchanged, worse" or "better" compared to the pre-injection status. An "unchanged" equals a transition score of 0. If the participant answers "worse", he/she is asked to rate the degree of worsening on a 7 point Likert scale, and the corresponding scores range from -1 to -7. Correspondingly, if a participant answers "better", he/she is asked to rate the degree of improvement on a 7 point Likert scale, and the corresponding scores range from 1 to 7. Thus the Transition score range from -7 (worsening) to 7 (improvement), with the mid-point - 0 - representing no change.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Study Protocol — http://www.parkerinst.dk